CLINICAL TRIAL: NCT06261567
Title: A Retrospective Chart Review to Investigate Clinical Remission in Patients With Severe Asthma Treated With Biologics in the United Kingdom National Health Service
Acronym: REMISSION UK
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00189
Record Dates: First submitted 2024-01-09; First posted 2024-02-15 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Biologic treatment — Patients receiving treatment with any biologic treatment for severe asthma which is approved within the UK NHS. These include omalizumab, mepolizumab, reslizumab, benralizumab and/or dupilumab

SUMMARY:
Asthma is a common lung condition that causes occasional breathing difficulties and affects around 5.4 million people in the UK of all ages. Common symptoms can include wheezing when breathing, breathlessness, a tight chest and coughing. However, these symptoms can get worse and lead to an asthma attack which can be fatal.

There is currently no cure for asthma but there are treatments that can help keep the symptoms under control. The main types of treatment include reliever inhalers used when needed quickly to reverse asthma symptoms for a short time, and preventer inhalers that are used everyday to prevent symptoms for starting. Unfortunately, not all patients are able to control their asthma on these treatments alone. Biologic treatments, also known as monoclonal antibodies, have been introduced to treat certain types of severe asthma over recent years. These specialist treatments use antibodies produced from cells in a laboratory to help reduce inflammation and might offer the possibility of higher levels of disease control including the reduction or absence of symptoms and normal lung function. This higher level of disease control is called remission.

This study aims to understand whether or not remission is possible in patients with severe asthmas treated with biologics in the NHS. This study will take place a 4 specialist asthma centres in the UK and seeks to include retrospective data from approximately 450 adult patients that were treated with biologics as part of routine care between 01 October 2021 and 30 September 2022. Data will be collected directly from medical records and entered into the study database in a pseudonymised format by members of the direct care team ready for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Initiated on a biologic treatment for SA between 1st October 2021 and 30th September 2022
* Patients who received ≥1 dose of biologic treatment
* Patients aged ≥18 years at index

Exclusion Criteria:

* Patients who were involved in any interventional clinical trial during the study period (+/- 12 months from index).

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population for this study will be patients who were treated with a biologic for severe asthma in UK NHS centres between October 2021 and September 2022
Sampling Method: Non-Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in clinical remission | 12 months
  Proportion of patients with zero exacerbations, zero mOCS use and ACQ <1.5
Number and proportion achieving specific criteria for clinical remission | 12 months
  Number and proportion achieving the following criteria for clinical remission:
  * any 1 criterion
  * any 2 criteria
  * any 3 criteria
  * exacerbation AND maintenance oral corticosteroids (mOCS) criteria
  * exacerbation, mOCS, AND asthma symptom control criteria
Number and proportion of super-responders | 12 months
Number and proportion of responders | 12 months
Number and proportion of non-responders | 12 months

SECONDARY OUTCOMES:
Age at index | Index (first dose of biologic)
Sex | Index (first dose of biologic)
Ethnicity | Index (first dose of biologic)
Smoking status | Index (first dose of biologic)
BMI | Index (first dose of biologic)
IMD quintile | Index (first dose of biologic)
Comorbidities | Index (first dose of biologic)
COVID-19 vaccination status | Index (first dose of biologic)
Fractional Exhaled Nitric Oxide (FeNO) | Index (first dose of biologic)
Blood eosinophil count (EOS) | Index (first dose of biologic)
IgE | Index (first dose of biologic)
ACQ-6 | Index (first dose of biologic)
AQLQ | Index (first dose of biologic)
lung function (FEV1) | Index (first dose of biologic)
Rate of exacerbation in prior 12 months | Index (first dose of biologic)
Asthma treatments at 6 months | 6 months
Asthma treatments at 12 months | 12 months
Annualised exacerbation rate (AER) | 6 months
mOCS use (proportion with 0 mg/day) | 6 months
ACQ-6 score | 6 months
AQLQ score | 6 months
Lung function (FEV-1) | 6 months
Respiratory infections | 6 months
Annualised exacerbation rate (AER) | 12 months
mOCS use (proportion with 0 mg/day) | 12 months
ACQ-6 score | 12 months
AQLQ score | 12 months
Lung function (FEV-1) | 12 months
Respiratory infections | 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Research Site, Birmingham
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2287R00189&attachmentIdentifier=cc2742bb-8af2-4172-aa01-b367bbd9edb8&fileName=D2287R00189_AZ_Remission_-_CSR_Synopsis_v0.1_24JULY2025.pdf&versionIdentifier=